CLINICAL TRIAL: NCT06419985
Title: A Phase 2 Single-arm, Open Label Clinical Trial to Evaluate the Efficacy of Ketamine HCl Prolonged Release Tablets in Participants With Complex Regional Pain Syndrome
Brief Title: Ketamine HCl Prolonged Release Oral Tablets for CRPS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Steven Richeimer, Professor of Clinical Anesthesiology, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23015-0001
Record Dates: First submitted 2024-05-06; First posted 2024-05-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Complex Regional Pain Syndromes
Keywords: CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 80mg Ketamine HCl PR (Experimental): One 40mg tablet of Ketamine HCl PR twice a day, which may be increased to two 40mg tablets Ketamine HCl PR twice a day at week 4 if subject does not experience adequate pain relief.
  Interventions: Drug: 80mg/day Ketamine HCl Prolonged Release; Drug: 160mg/day Ketamine HCl Prolonged Release

INTERVENTIONS:
Drug: 80mg/day Ketamine HCl Prolonged Release — Administration of Ketamine HCl Prolonged Release - 40mg BID
  Other Names: 80mg Ketamine PR
Drug: 160mg/day Ketamine HCl Prolonged Release — Administration of Ketamine HCl Prolonged Release - 80mg BID
  Other Names: 160mg Ketamine PR

SUMMARY:
The purpose of this study is to evaluate the efficacy of Ketamine HCl Prolonged Release (PR) tablets in participants with pain due to complex regional pain syndrome (CRPS).

Additionally, this trial will explore the feasibility of the trial design through dosing compliance, clinical instruments for safety and quality of life measurements, and pharmacokinetic profile.

DETAILED DESCRIPTION:
This study will enroll patients (age 18 to 64 years old) with history of CRPS (diagnosis greater than 6 months prior) at a single academic medical institution in the United States. All participants will be informed about the study and potential risks and will provided written informed consents prior to undergoing any study-related procedures.

Health status assessments including physical exams, blood work, urinalysis, EKG and questionnaires to assess quality of life and pain scale measurement will be conducted at the clinic visits. The participants will also keep a daily diary throughout the study to record pain levels, daily blood pressure and any additional pain medication needed.

There will be a total of 10 visits: a screening visit (day -28 to -7), clinic visits at day 1 (Baseline), week 2, week 4, week 8, and at the end of study (EOS) visit at 12 weeks. There will be additional telemedicine visits at week 1, week 3, week 5 and at the safety followup visit approximately 4 weeks after the EOS visit. There will also be followup phone call throughout the study to check on compliance and any adverse events.

All subjects will start with 40mg BID of Ketamine PR (80 mg/day) on the Baseline visit. The subjects are required to be observed in person for 6 hours following the first dose for any side effects using the Ketamine Side Effects Tools (KSET) - Baseline and Acute Treatment forms [From: Brooke Short et al. "Development of ketamine side effect tool (KSET) as a reference: J Affect Disord. 2020 April 01; 266: 615-620. doi:10.1016/j.jad.2020.01.120].

At an in person clinic visit 4 weeks after the Baseline visit, the dose may be increased to 80 mg BID (160 mg/day), using the same observation period as described at the Baseline visit. The study drug dosage will only be increased at this visit if the subject has not experienced adequate pain relief and has not experienced any adverse events.

Administration of the study drug will stop at the EOS visit (at 12 weeks after the Baseline visit).

Hemodynamic measurements, laboratory results, KSET - Followup form results and examination by the PI/Co-PI will be used throughout the study to assess possible adverse events (AEs). If the subject experiences any Grade 2 AEs, the PI/Co-PI will use clinical expertise and best judgement after determining the subject's level of distress and or discomfort to decide whether the subject will remain at the current dose, decrease the dose or discontinue study drug. If the subject experiences any Grade 3 Adverse Events (AEs), the study drug will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants between 18 and 64 years of age, inclusive, at Screening Visit.
2. Participants with a documented history of CRPS of at least 6 months at Visit 1.
3. At least one sign in two of the categories of The Budapest Criteria for CRPS to support the diagnosis of CRPS.
4. Stable individual regular standard treatment regimen for CRPS pain, i.e., no change in drug and non-drug treatments for at least 4 weeks prior to Screening Visit and anticipated to remain stable throughout the study.
5. No surgery, denervation procedures or neural blockade within 1 month of Screening Visit.
6. Participants on ketamine therapy at Screening Visit must agree to discontinue use for at least 14 days prior to the Baseline Observation Period.
7. Agree to discontinue any prohibited medications within prior to 14 days of the Baseline Observation Period and for the duration of the study.
8. Average daily CRPS pain intensity score in the affected limb of ≥5 and ≤9 on an 11-point (0-10) NRS averaged over 7 days prior to Baseline Visit (Visit 1). This will be based on completion of at least 5 daily pain diary entries during the week prior to Visit 1, with no more than one 24-hour pain intensity score of zero or more than one 24-hour pain intensity score of 10.
9. Participants willing and able (e.g., mental and physical condition) to participate in all aspects of the trial, including use of medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements as evidenced by providing signed written informed consent at Screening Visit.
10. For persons of reproductive potential: use of highly effective contraception (females: barrier (condom, diaphragm, sponge, cervical cap) and/or oral, implantable rod, or intrauterine device birth control; males: barrier (condom)) for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 weeks after the end of study intervention administration.

Exclusion Criteria:

1. Known or suspected cardiovascular disease, arrythmias, and/or respiratory issues.
2. Abnormal EKG results, abnormal blood pressure (SBP <90 or ≥ 140; DBP <50 or ≥ 90) and/or heart rates (<50 or >110).
3. Known or suspected psychotic illness or neurologic disease.
4. Known or suspected elevated intraocular and/or intracranial pressure.
5. Known or suspected renal or urologic conditions or symptoms (i.e., bladder pain syndrome, interstitial cystitis), and/or abnormal baseline urinalysis results.
6. Known or suspected hyperthyroidism.
7. Allergy, hypersensitivity, or intolerance to ketamine or any of the investigational product excipients.
8. Participants receiving opioids ≥30 mg/day morphine milligram equivalents (MME), whether as part of their individual standard treatment regimen for CRPS pain or in context with any other indication, within the last two weeks prior to Visit 1.
9. Positive urine screen for any of the following: cocaine, amphetamine, methamphetamine, PCP, opioids, THC (other than medication used for individual standard treatment of pain) at Visit 1.
10. Known or suspected acute or chronic alcoholism, delirium tremens, or toxic psychosis.
11. Meet DSM-5 criteria for current or past substance use disorder within the last 5 years for any psychoactive substances other than nicotine or caffeine.
12. Known hepatic dysfunction or serious liver disease, including presence of aspartate aminotransferase (AST) levels ≥ 2 X upper limit of normal and/or alanine aminotransferase (ALT) levels ≥ 2 X upper limit of normal and/or total bilirubin ≥ 1.5 X upper limit of normal
13. Abnormal urinalysis, urine culture or abnormal creatinine
14. Evidence of moderate or severe renal impairment (CRCL <60 ml/min) or participants with renal failure who are on any form of dialysis.
15. Current or previous history of seizures.
16. A positive pregnancy test/confirmed pregnancy test at the screening or baseline visit.
17. If Ask Suicide-Screening Questionnaire (ASQ) is positive at Grade 2 (moderate), subject will be excluded.
18. Any other condition of the patient that in the opinion of the investigator may compromise evaluation of the trial treatment or may jeopardize participant's safety, compliance or adherence to protocol requirements.
19. Previous enrollment in this trial or participation in any other clinical trial within the past 30 days prior to enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Average Daily Pain Numerical Rating Scale (ADP NRS) | Day 1 to week 12
  Average Daily Pain Numerical Rating Scale is a validated, self-reported instrument used to assess average pain intensity level over the past 24 hours. It uses an 11-point (0-10) scale, with 0 being "no pain" and 10 being "worst pain imaginable."

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System-2 (PROMIS-29 Profile v2.1) | Day 1 to week 12
  The PROMIS-29 Profile v2.1 is a validated, self-reported instrument to measure functioning and well-being in 7 categories: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities and pain interference. There are 4 questions in each of the 7 categories. Each question has five responses with a score from 1 to 5 (1 being best and 5 being worst). For each of these 7 categories, the lowest score is 4; the highest is 20.
Complex Regional Pain Syndrome Severity Scale (CSS) | Day 1 to week 12
  The CSS Questionnaire assesses changes in Complex Regional Pain Syndrome (CRPS) severity by asking for the presence or absence (score of 1 or 0) of 16 clinically assessed signs and symptoms of CRPS. A higher score is worse, indicate greater CRPS severity (range 0-16).
Patient Global Impression of Change (PGIC) | Day 1 to week 12
  Patient Global Impression of Change is a validated, self-reported instrument consisting of a 7-point scale (1 through 7) depicting a patient's rating of overall improvement since a certain point in time. The higher PGIC scores, the greater improvement. We will compare the scores at the end of Cycle 1 (1-4 weeks), 2 (4-8 weeks), and 3 (8-12 weeks).
Maximum Plasma concentration [Cmax] of Ketamine | Day 1 to Day 7
  Maximum Plasma concentration [Cmax] is the maximum concentration of the drug, Ketamine, in the body, measured in grams/Liter. Blood samples are obtained at Day 2, 4, and 7.
Time to Maximum Plasma concentration [Tmax] of Ketamine | Day 1 to Day 7
  Time to Maximum Plasma concentration [Tmax] is the time it takes for the drug Ketamine, to reach maximum concentration (Cmax), measured in minutes. Blood samples are obtained at Day 2, 4, and 7.
Opioid sparing | Day 1 to week 12
  Participants will record any change in the amount (expressed as MME) and frequency of opioid medications used for treating CRPS pain.
Medication sparing | Day 1 to week 12
  Participants will record daily use of rescue medication (expressed in mg and number of tablets) for treating CRPS pain. Acetaminophen (up to 3000mg/day) will be offered as rescue medication for breakthrough pain.
Safety of Ketamine HCl PR oral tablets | Day 1 to 18 weeks
  Number of participants with AEs, with abnormal vital signs, abnormal physical examination parameters; abnormal Electrocardiogram (EKG) parameters; abnormal laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Steven Richeimer, MD, Principal Investigator — Keck Medical Center of USC
Locations (1):
- Pain Center, Keck Medical Center of University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sammy Al Mukhaizeem, et al. Investigating the effectiveness of oral ketamine on pain, mood and quality of life in treatment resistant chronic pain — http://DOI.org/10.3389/fpain.2023.1268985
- See also: Megan Dutton, et al. Oral ketamine may offer a solution to the ketamine conundrum — https://doi.org/10.1007/s00213-023-06480-x
- See also: Mark C. Enarson, et al. Clinical Experience with Oral Ketamine — https://pubmed.ncbi.nlm.nih.gov/10355218/
- See also: Glue, et al. Extended-release ketamine tablets for treatment-resistant depression: A randomized placebo-controlled phase 2 trial — https://doi.org/10.1038/s41591-024-03063-x
- See also: Hasan, M. et al. Chiral Pharmacokinetics and Metabolite Profile of Prolonged-release Ketamine Tablets in Healthy Human Subjects — https://doi.org/10.1097/ALN.0000000000003829
- See also: Naim Zaki, et al. Long-term safety and maintenance of response with esketamine nasal spray in participants with treatment-resistant depression: interim results of the SUSTAIN-3 study — https://doi.org/10.1038/s41386-023-01577-5